CLINICAL TRIAL: NCT01944722
Title: Clinical Evaluation of the BD Onclarity™ HPV Assay on the BD Viper™ LT System With Cervical Specimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BDS-USHPV
Record Dates: First submitted 2013-09-05; First posted 2013-09-18 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BD Onclarity™ HPV assay on BD Viper™ LT (Experimental): The LBC specimen will be tested with the BD Onclarity™ HPV assay on the BD Viper™ LT instrument. Colposcopy will be performed on subjects who have abnormal cytology or HPV positive test results or from a random sampling of subjects with normal cytology and HPV negative test results.
  Interventions: Device: BD Onclarity™ HPV assay on BD Viper™ LT; Procedure: Colposcopy

INTERVENTIONS:
Device: BD Onclarity™ HPV assay on BD Viper™ LT — The BD HPV specimen will be tested with the BD Onclarity™ HPV assay on the BD Viper™ LT instrument. The results will be compared to adjudicated histology. A portion of the specimens will be compared to a composite comparator generated by results of both Digene HPV and a polymerase chain reaction (PCR) sequencing test.
Procedure: Colposcopy — Colposcopy will be performed on subjects that have abnormal cytology or HPV positive test results or random sampling of subject with normal cytology and HPV negative test results.

SUMMARY:
The purpose of the study is to compare the results of the Becton Dickinson (BD) Onclarity™ Human Papilloma Virus (HPV) Assay on the BD Viper™ LT instrument from liquid-based cytology (LBC) media diluted in BD HPV LBC diluent to adjudicated histology results from biopsy and a molecular composite comparator.

ELIGIBILITY:
Inclusion Criteria:

* Females who are >21 years of age
* Females who provide informed consent

Exclusion Criteria:

* Known pregnant
* Cervical cytology specimen collected within the last 4 months
* Prior complete or partial hysterectomy involving removal of cervix
* Application of chemical compounds to the cervical area 24 hour prior to study entry- acetic acid, iodine, spermicide, douche, or anti-fungal medications
* Conization, Loop Electrosurgical Excision Procedure (LEEP), cervical laser surgery or cryosurgery on the cervix has been performed in the last twelve months
* Enrolled in a cervical disease diagnostic trial since 2007.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33858 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cooper, MD, Study Director — Becton, Dickinson and Company
Locations (41):
- United States (41):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Mobile OB/GYN, Mobile, Alabama
  - Women's Health Research of Arizona, Phoenix, Arizona
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Women's Health Care Research Corp, San Diego, California
  - West Coast Medical Research, San Diego, California
  - Blueskies Center for Women, Colorado Springs, Colorado
  - Health Awareness Inc, Jupiter, Florida
  - Altus, Lake Worth, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Medical Network for Education and Research, Decatur, Georgia
  - Fellows Research Associates - Savannah, Savannah, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Indiana University, Indianapolis, Indiana
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Louisiana State University, New Orleans, Louisiana
  - Saginaw Valley Medical Research, Saginaw, Michigan
  - Transgenomics, Omaha, Nebraska
  - Vitura / Phoenix, Moorestown, New Jersey
  - Meridian Health, Neptune City, New Jersey
  - Q Squared Solutions, Teterboro, New Jersey
  - TriCore Reference Laboratory, Albuquerque, New Mexico
  - Research Pathology Associates, LLC, Irvington, New York
  - Montefiore Medical Center, The Bronx, New York
  - LabCorp, Burlington, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - HWC Women's Research Center, Englewood, Ohio
  - Center for Women's Health of Lansdale, Lansdale, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Reading Health Physicians Network, West Reading, Pennsylvania
  - Fellows Research Associates - Bluffton, Bluffton, South Carolina
  - James T Martin Jr, MD, North Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Center for Disease Detection (CDD), San Antonio, Texas
  - Physicians Research Options, Draper, Utah
  - Research Pathology Associates, Earlysville, Virginia
  - Tidewater Clinical, Virginia Beach, Virginia

REFERENCES:
- [Derived] Stoler MH, Wright TC, Parvu V, Yanson K, Eckert K, Kodsi S, Cooper C. HPV Testing With 16, 18, and 45 Genotyping Stratifies Cancer Risk for Women With Normal Cytology. Am J Clin Pathol. 2019 Mar 1;151(4):433-442. doi: 10.1093/ajcp/aqy169. PMID 30649177
- [Derived] Wright TC Jr, Stoler MH, Parvu V, Yanson K, Eckert K, Kodsi S, Cooper CK. Detection of Cervical Neoplasia by Human Papillomavirus Testing in an Atypical Squamous Cells-Undetermined Significance Population: Results of the Becton Dickinson Onclarity Trial. Am J Clin Pathol. 2019 Jan 1;151(1):53-62. doi: 10.1093/ajcp/aqy084. PMID 30189049
- [Derived] Stoler MH, Wright TC Jr, Parvu V, Vaughan L, Yanson K, Eckert K, Karchmer T, Kodsi S, Cooper CK. The Onclarity Human Papillomavirus Trial: Design, methods, and baseline results. Gynecol Oncol. 2018 Jun;149(3):498-505. doi: 10.1016/j.ygyno.2018.04.007. Epub 2018 Apr 19. PMID 29681462

RESULTS

PARTICIPANT FLOW:
Groups:
- BD Onclarity™ HPV Assay on BD Viper™ LT: The LBC specimen will be tested with the BD Onclarity™ HPV assay on the BD Viper™ LT instrument. The results will be compared to adjudicated histology. A portion of the specimens will be compared to a composite comparator generated by results of both Digene (HC2) HPV and a polymerase chain reaction (PCR) sequencing test.
  Colposcopy will be performed on subjects that have abnormal cytology or HPV positive test results or a random sampling of subjects with normal cytology and HPV negative test results.
Period: Overall Study
Arm/Group | BD Onclarity™ HPV Assay on BD Viper™ LT
Started | 33858
Completed | 24343
Not Completed | 9515
Not completed — Didn't meet Inclusion/Exclusion Criteria | 171
Not completed — Specimen Shipping Issues | 34
Not completed — Improper Storage/Transport | 5
Not completed — Insufficient Volume for Test | 1
Not completed — Missing Specimens | 3
Not completed — Specimens Mislabeled | 2
Not completed — Withdrawal by Subject | 8
Not completed — NILM Subjects <30 years old | 8106
Not completed — Unsatisfactory Cytology Result | 63
Not completed — >ASCUS Cytology | 1122

BASELINE CHARACTERISTICS:
Groups:
- ASCUS Aged 21 Years and Older: Participants aged 21 years and older and having atypical squamous cells of undetermined significance (ASCUS).
- NILM Aged 30 Years and Older: Participants aged 30 years and older and having cytology results that are negative for intraepithelial lesions or malignancy (NILM).
- Total: Total of all reporting groups
Arm/Group | ASCUS Aged 21 Years and Older | NILM Aged 30 Years and Older | Total
Number analyzed (Participants) | 1960 | 22383 | 24343
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (11.5) | 43.9 (9.6) | 43.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1960 | 22383 | 24343
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 303 | 4592 | 4895
  Not Hispanic or Latino | 1657 | 17789 | 19446
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 97 | 104
  Asian | 20 | 336 | 356
  Native Hawaiian or Other Pacific Islander | 4 | 60 | 64
  Black or African American | 459 | 3722 | 4181
  White | 1446 | 17988 | 19434
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 180 | 204
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1960 | 22383 | 24343

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the BD Onclarity™ HPV Assay for the Detection Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN)2 or Greater
Description: Sensitivity is calculated: Number of subjects with a positive BD Onclarity™ HPV test with adjudicated histology results of CIN2 or greater divided by the total number of subjects with adjudicated histology results of CIN2 or greater (multiplied by 100).
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ASCUS >= 21 Years Old: Participants aged 21 years and older and having atypical squamous cells of undetermined significance (ASCUS)
- NILM >= 30 Years Old: Participants aged 30 years and older and having cytology results negative for intraepithelial lesions or malignancy
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants | 85.7 [77.8 to 91.1] | 44.4 [27.7 to 76.2]

2. Primary Outcome: Sensitivity of the BD Onclarity™ HPV Assay for the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN)3 or Greater
Description: Sensitivity is calculated: Number of subjects with a positive BD Onclarity™ HPV test with adjudicated histology results of CIN3 or greater divided by the total number of subjects with adjudicated histology results of CIN3 or greater (multiplied by 100).
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NILM >= 30 Years Old | ASCUS >= 21 Years Old
Number analyzed (Participants) | 22383 | 1960
percentage of participants | 69.3 [42.0 to 100.0] | 91.4 [77.6 to 97.0]

3. Primary Outcome: Specificity of the BD Onclarity™ HPV Assay for Detecting Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN)2 or Greater
Description: Specificity is calculated: Number of subjects with a negative BD Onclarity™ HPV test with adjudicated histology results of CIN2 or greater divided by the total number of subjects with adjudicated histology results of less than CIN2 (multiplied by 100).
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants | 64.1 [61.7 to 66.5] | 92.4 [92.1 to 92.8]

4. Primary Outcome: Specificity of the BD Onclarity™ HPV Assay for Detecting Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN)3 or Greater
Description: Specificity is calculated: Number of subjects with a negative BD Onclarity™ HPV test with adjudicated histology results of CIN3 or greater divided by the total number of subjects with adjudicated histology results of less than CIN3 (multiplied by 100).
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants | 62.0 [59.6 to 64.4] | 92.3 [92.0 to 92.7]

5. Primary Outcome: Positive Predictive Value (PPV) of the BD Onclarity™ HPV Assay for Detecting Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN).
Description: Positive Predictive Value is calculated: Number of subjects with a positive result for the BD Onclarity™ HPV test and adjudicated histology results of CIN2 or greater divided by the total number of subjects with positive result for the BD Onclarity™ HPV test (multiplied by 100). Similar for CIN3 or greater.
Time Frame: Up to 14 weeks
Population: Data includes all participants with evaluable data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants
  CIN2 or greater | 14.3 [13.0 to 15.5] | 5.1 [3.9 to 6.3]
  CIN3 or greater | 5.1 [4.3 to 5.6] | 3.0 [2.1 to 3.9]

6. Primary Outcome: Negative Predictive Value (NPV) of the BD Onclarity™ HPV Assay for Detecting Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN).
Description: Negative Predictive Value is calculated: Number of subjects with a negative result for the BD Onclarity™ HPV test and histology results less than CIN2 divided by the total number of subjects with negative results for the BD Onclarity™ HPV test (multiplied by 100). Similar for CIN3 or greater.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants
  CIN2 or greater | 98.5 [97.6 to 99.0] | 99.5 [99.0 to 99.9]
  CIN3 or greater | 99.7 [99.2 to 99.9] | 99.9 [99.7 to 100.0]

7. Primary Outcome: Likelihood Ratio for the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN2 or Greater).
Description: The likelihood ratio for each BD Onclarity™ HPV test outcome summarizes how many times more (or less) likely subjects with CIN2 or greater disease are to have that particular BD HPV Onclarity™ test outcome than subjects without the disease. Significant likelihood ratios (defined in cases where 1 is not contained within the 95% confidence interval) indicate that a test result is informative.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
Ratio
  HPV High Risk Positive | 2.39 [2.13 to 2.63] | 5.86 [3.63 to 10.11]
  HPV 16 Positive | 5.98 [4.15 to 8.42] | 11.27 [5.92 to 21.08]
  HPV 18 Positive | 2.86 [1.24 to 6.45] | 4.41 [0 to 11.90]
  HPV 45 Positive | 1.16 [0.38 to 3.42] | 2.42 [0 to 7.18]
  HPV 16/18/45 Positive | 4.12 [3.07 to 5.38] | 8.06 [4.48 to 14.46]
  11 Other High Risk HPV Positive | 1.75 [1.38 to 2.15] | 4.92 [3.0 to 8.51]
  HPV High Risk Negative | 0.22 [0.14 to 0.35] | 0.6 [0.26 to 0.78]

8. Primary Outcome: Likelihood Ratio for the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN3 or Greater).
Description: The likelihood ratio for each BD Onclarity™ HPV test outcome summarizes how many times more (or less) likely subjects with CIN3 or greater disease are to have that particular BD Onclarity™ HPV test outcome than subjects without the disease. Significant likelihood ratios (defined in cases where 1 is not contained within the 95% confidence interval) indicate that a test result is informative.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
Ratio
  HPV High Risk Positive | 2.41 [2.03 to 2.64] | 9.02 [5.48 to 13.21]
  HPV 16 Positive | 8.6 [5.69 to 12.08] | 21.42 [11.10 to 38.33]
  HPV 18 Positive | 1.28 [0.22 to 6.74] | 7.64 [0 to 22.64]
  HPV 45 Positive | 1.15 [0.20 to 6.03] | 3.16 [0 to 12.28]
  HPV 16/18/45 Positive | 5.35 [3.72 to 7.07] | 14.92 [8.19 to 25.88]
  11 Other High Risk HPV Positive | 1.26 [0.76 to 1.88] | 6.49 [3.59 to 10.98]
  HPV High Risk Negative | 0.14 [0.05 to 0.36] | 0.33 [0 to 0.63]

9. Primary Outcome: Absolute Risk for the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN2 or Greater).
Description: The Absolute Risk (AR) of CIN2 or greater disease for each BD Onclarity™ HPV test outcome is the probability of the disease for that particular BD Onclarity™ HPV test outcome. A higher absolute risk indicates a higher probability overall for an event to occur.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of assays
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of assays
  HPV High Risk Positive | 14.3 [13.0 to 15.5] | 5.1 [3.9 to 6.3]
  HPV 16 Positive | 29.5 [22.5 to 37.0] | 9.3 [5.5 to 13.7]
  HPV 18 Positive | 16.7 [7.9 to 31.1] | 3.9 [0.0 to 8.4]
  HPV 45 Positive | 7.5 [2.6 to 19.3] | 2.2 [0.0 to 5.4]
  HPV 16/18/45 Positive | 22.3 [17.7 to 27.3] | 6.8 [4.4 to 9.7]
  11 Other High Risk HPV Positive | 10.9 [8.8 to 13.1] | 4.3 [3.1 to 5.5]
  HPV High Risk Negative | 1.5 [1.0 to 2.4] | 0.5 [0.1 to 1.0]

10. Primary Outcome: Absolute Risk for the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN3 or Greater).
Description: The Absolute Risk (AR) of CIN3 or greater disease for each BD Onclarity™ HPV test outcome is the probability of the disease for that particular BD Onclarity™ HPV test outcome. A higher absolute risk indicates a higher probability overall for an event to occur.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of assays
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of assays
  HPV High Risk Positive | 5.1 [4.3 to 5.6] | 3.0 [2.1 to 3.9]
  HPV 16 Positive | 16.1 [11.2 to 21.2] | 6.9 [3.9 to 9.9]
  HPV 18 Positive | 2.8 [0.5 to 13.0] | 2.6 [0.0 to 6.4]
  HPV 45 Positive | 2.5 [0.4 to 11.8] | 1.1 [0.2 to 3.4]
  HPV 16/18/45 Positive | 10.6 [7.7 to 13.6] | 4.9 [3.0 to 6.9]
  11 Other High Risk HPV Positive | 2.7 [1.7 to 4.0] | 2.2 [1.4 to 3.2]
  HPV High Risk Negative | 0.3 [0.1 to 0.8] | 0.1 [0.0 to 0.3]

11. Primary Outcome: Relative Risk of the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN2 or Greater).
Description: Relative Risk is the ratio between two different absolute risks. The relative risk of having CIN2 or greater disease will be evaluated to compare two different BD Onclarity™ HPV Assay test outcomes.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
ratio
  HPV HR Positive vs HPV HR Negative | 9.33 [5.49 to 15.88] | 9.31 [4.5 to 38.03]
  HPV 16/18/45 Positive vs HPV HR Negative | 14.57 [8.3 to 25.52] | 12.56 [5.62 to 49.57]
  HPV 16/18/45 Positive vs 11 Other HR HPV Positive | 2.05 [1.41 to 2.98] | 1.59 [0.97 to 2.57]
  11 Other HR HPV Positive vs HPV HR Negative | 7.1 [4.05 to 12.45] | 7.88 [3.81 to 32.06]

12. Primary Outcome: Relative Risk of the Detection of Cervical Disease as Defined by Cervical Intraepithelial Neoplasia (CIN3 or Greater).
Description: Relative Risk is the ratio between two different absolute risks. The relative risk of having CIN3 or greater disease will be evaluated to compare two different BD Onclarity™ HPV Assay test outcomes.
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
ratio
  HPV HR Positive vs HPV HR Negative | 16.59 [5.42 to 50.86] | 26.36 [8.51 to 9999999]
  HPV 16/18/45 Positive vs HPV HR Negative | 34.68 [11.09 to 108.53] | 42.78 [13.16 to 9999999]
  HPV 16/18/45 Positive vs 11 Other HR HPV Positive | 3.91 [1.98 to 7.73] | 2.24 [1.22 to 4.05]
  11 Other HR HPV Positive vs HPV HR Negative | 8.87 [2.70 to 29.14] | 19.14 [5.83 to 9999999]

13. Primary Outcome: Positive Percent Agreement of the BD Onclarity™ HPV Assay as Compared to a Composite HPV Comparator Incorporating Results for the Digene Hybrid Capture 2 (HC2) HPV Test and PCR/Sequencing on Both Strands of the PCR Amplicon (Bidirectional Sequencing)
Description: Positive percent agreement is calculated: Number of subjects with a positive BD Onclarity™ HPV test with composite comparator positive divided by the total number of subjects with composite comparator positive (multiplied by 100).
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants | 97.4 [95.5 to 98.6] | 92.0 [89.8 to 94.0]

14. Primary Outcome: Negative Percent Agreement of the BD Onclarity™ HPV Assay Compared to a Composite HPV Comparator Incorporating Results for the Digene HC2 HPV Test and PCR/Sequencing on Both Strands of the PCR Amplicon (Bidirectional Sequencing)
Description: Negative percent agreement is calculated: Number of subjects with a negative BD Onclarity™ HPV test with composite comparator negative divided by the total number of subjects with composite comparator negative (multiplied by 100).
Time Frame: Up to 14 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
percentage of participants | 98.5 [97.1 to 99.2] | 99.4 [99.3 to 99.6]

15. Primary Outcome: Non-reportable Rate of the BD Onclarity™ HPV Test
Description: Non-reportable rate is calculated as the number of non-reportable BD Onclarity™ HPV test results divided by the total number of BD Onclarity™ HPV test results (multiplied by 100). Not included in this calculation are specimens that did not yield a result due to specimen labeling, processing and volume issues.
Time Frame: Up to 14 weeks
Measure: Number; unit: percentage of participants
Arm/Group | BD Onclarity™ HPV Assay on BD Viper™ LT
Number analyzed (Participants) | 33570
percentage of participants | 0.24

16. Primary Outcome: Number of Participants With Cervical Intraepithelial Neoplasia (CIN)2 or Greater and CIN3 or Greater Within Each Cytology Category.
Description: Prevalence is calculated as the rate of CIN2 or greater and CIN3 or greater within each cytology category.
Time Frame: Up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ASCUS >= 21 Years Old | NILM >= 30 Years Old
Number analyzed (Participants) | 1960 | 22383
Participants
  CIN2 or greater | 105 | 80
  CIN3 or greater | 35 | 46

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the course of the study (up to 30 months).
Groups:
- BD HPV Onclarity™ Assay on BD Viper™ LT: Subjects tested with the BD HPV Onclarity™ assay on the BD Viper™ LT instrument.
Arm/Group | BD HPV Onclarity™ Assay on BD Viper™ LT
All-Cause Mortality (participants affected / at risk) | 2/33858
Serious Adverse Events (participants affected / at risk) | 9/33858
Other Adverse Events (participants affected / at risk) | 0/33858
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BD HPV Onclarity™ Assay on BD Viper™ LT (N=33858)
Diverticultitis and Sepsis (Infections and infestations) | 1 (1)
Squamous cell carcinoma in situ - cervical (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myomectomy (Surgical and medical procedures) | 1 (1)
Prescription overdose leading to death (Injury, poisoning and procedural complications) | 1 (1)
Stage 3 Breast Infiltrating Ductal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary Thyroid Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma of vulva, in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Right Breast Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes